CLINICAL TRIAL: NCT01766115
Title: Hepatitis C Virus Post-Exposure Prophylaxis for Health Care Workers
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Raymond T. Chung, MD, Director of Hepatology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2012P000954
Record Dates: First submitted 2013-01-07; First posted 2013-01-11 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Viral Hepatitis C
Keywords: HCV; needlestick; occupational; transmission; health care worker; telaprevir
MeSH Terms: conditions — Hepatitis C; Needlestick Injuries | interventions — telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Telaprevir (Experimental): 750 mg oral tablet of telaprevir will be given three times per day for 4 weeks within a five (5) day period from health care worker exposure.
  Interventions: Drug: Telaprevir

INTERVENTIONS:
Drug: Telaprevir — HCV Protease Inhibitor
  Other Names: Incivek

SUMMARY:
To assess the safety and tolerability of the use of telaprevir in the setting of post-exposure prophylaxis among HCW exposed to HCV genotype 1 or genotype 2.

To assess the election rate of postexposure prophylaxis for HCV-related occupational exposures in HCW.

DETAILED DESCRIPTION:
At MGH and BWH, HCW exposed to blood or visibly bloody fluids are referred immediately to Occupational Health Services. The person whose blood or body fluid is the source of an occupational exposure should be evaluated for HBV, HCV, and HIV infection. Information available in the medical record at the time of exposure, or from the source person, might confirm or exclude bloodborne virus infection. If the HBV, HCV, and/or HIV infection status of the source is unknown, the source patient should be informed of the incident and tested for serologic evidence of bloodborne virus infection, including HBsAg, HCV antibody, and HIV antibody. Reactive results by EIA for anti-HCV are confirmed by HCV RNA PCR, which is tested using Roche COBAS TaqMan quantitative assay (Roche Molecular Systems) with a lower limit of quantitation of < 43 IU/ml. HCV RNA testing is performed twice weekly at MGH and BWH. In the event that the source patient's HCV antibody is positive and the HCV RNA is below the lower limit of detection, an HCV Recombinant Immunoblot Assay (RIBA) will be ordered: if the RIBA is negative, then the positive HCV antibody is interpreted as a false positive result, and the source patient is not infected with HCV. If the RIBA is positive, the source patient will then receive serial HCV RNA testing

For HCW exposed to an HCV-positive source, HCV antibody testing is performed at the time of exposure. Per standard practices recommended by Partners Occupational Health Services, HCV RNA testing of HCW is not performed at the time of exposure, unless the HCV antibody test is positive. For the current study, if a HCW meets inclusion criteria (specifically, has an exposure through needlestick injury with a hollow-bore needle to a source patient who is anti-HCV(+) and HCV RNA (+); and the HCW is anti-HCV Ab negative) and is interested in enrolling in the study, HCV RNA testing of eligible HCW will be performed at the initial visit.

For potential study enrollment, patients will be directly referred from Partners Occupational Health Services (BWH or MGH). They will be responsible for contacting study personnel by pager. In the event that the exposure occurs after the Occupational Health Services office is closed, the HCW will be evaluated in the Emergency Room as per standard protocol, and will be referred to study personnel the following business day. The HCW will then be screened with an interview in person, and patients with an appropriate exposure will be eligible for inclusion.

Study drug will be offered to subjects who were exposed to potentially HCV-infected blood after needlestick injury with hollow-bore needles. Blood on intact skin is considered low-risk and, therefore, treatment will not be recommended. Other unusual injuries/exposures will be included on an individual basis by study physicians.

Once the HCW signs informed consent to participate in the study, he/she will be offered a prescription for PEP with telaprevir 750 mg three times per day for 4 weeks within a five (5) day period from his/her exposure.

Telaprevir has been shown to interact with both HIV protease inhibitors and reverse transcriptase inhibitors through their activity upon the CYP3A enzyme. With respect to the interactions between telaprevir and HIV protease inhibitors, it is not recommended to co-administer darunavir/ritonavir, fosamprenavir/ritonavir, or lopinavir/ritonavir with telaprevir[19]. In addition, regarding the use of reverse transcriptase inhibitors, concomitant administration of telaprevir and efavirenz resulted in reduced steady-state exposures to telaprevir and efavirenz. Van Heeswijk et al conducted three open-label, randomized cross-over trials among HIV and HCV negative healthy volunteers, and found that therapeutic levels of telaprevir, efavirenz, and tenofovir were maintained when the telaprevir dose was increased to 1250 mg three-times daily.

As a result of these interactions, in cases where a HCW is exposed to HCV and HIV and elects to take HIV PEP, telaprevir will be offered for HCV PEP if one of the following HIV PEP regimens is prescribed:

1. Tenofovir/Emtricitabine (Truvada) + Atazanavir/Ritonavir
2. Tenofovir/Emtricitabine (Truvada) + Raltegravir

All decisions regarding post-exposure prophylaxis for HCW exposed to HCV and HIV will be discussed with the HIV/ID fellow.

Furthermore, for HCW who are HIV-infected and receiving HAART at the time of study enrollment, discussions will be held between the study team and the Infectious Disease specialist who is managing the HAART regimen of the HCW, in order to determine whether the patient could safely take telaprevir for HCV PEP.

The HCW will have anti-HCV testing performed, along with stored serum for lookbacks if necessary, as is the current protocol in Occupational Health. In addition to the usual laboratories drawn by occupational health (HCV antibody at week 0, HCV RNA at weeks 4 and 12), a blood count including differential will be required prior to consideration of study drug.

At week 4, all enrolled patients will have quantitative HCV viral load testing (regardless of treatment election). If HCV RNA is detectable, HCW will be referred to GI/Hepatology for consideration of intensified antiviral therapy. If negative for patients in the treatment arm, then telaprevir will be discontinued at this time.

At week 12 and 24, HCV RNA testing will be repeated. If positive, the patient will be referred for intensified antiviral therapy. Week 24 HCV RNA testing is necessary to look for the possibility that early prophylaxis with telaprevir delays the onset of hepatitis C infection.

ELIGIBILITY:
Inclusion Criteria:

* MGH or BWH health care workers with exposure through needlestick injury with hollow-bore needles to source patients who are anti-HCV (+) and HCV RNA (+)
* HCW is anti-HCV Ab negative. HCW exposed through needlestick injury with hollow-bore needles to source patients who are anti-HCV (+) and HCV RNA (-), regardless of the RIBA result, will not be eligible for the study. In addition, efforts will be made to identify the source patient's genotype, and if the genotype is unknown, then genotype testing will be performed. If the genotype is 2 or 3, then the HCW exposed to the source patient will not be eligible for the study.
* HCW will be eligible if exposed to a source patient who has a genotype 1, or if the genotype of the source patient is unknown or unable to be ascertained

Exclusion Criteria:

* Exposure to patient with known HCV genotype 2 or 3
* HCV Ab positive
* HCV Ab negative and HCV RNA > 1000 IU/ml
* Active malignancy
* Other condition in the opinion of the investigators or occupational health that makes telaprevir contraindicated in HCW
* Subjects with pre-existing end stage renal impairment or severe hepatic impairment (Child Pugh B or C), and anemia (starting hemoglobin 10 or less) will be excluded.
* Pregnant women will be excluded from the study. All female participants with reproductive potential will undergo a pregnancy test (specifically qualitative urine human chorionic gonadotropin), and those who test positive will not be eligible for study inclusion. Women whom are not pregnant and elect to enroll in the study will be advised that hormonal contraceptives may not be reliable during the study period and for up to two weeks following cessation of the study drug. During this time, female patients of childbearing potential should use two non-hormonal methods of effective birth control, examples of which include a male condom with spermicidal jelly OR female condom with spermicidal jelly (a combination of a male condom and a female condom is not suitable), a diaphragm with spermicidal jelly, a cervical cap with spermicidal jelly, or an intrauterine device (IUD).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | One year
  We seek to monitor the safety and tolerability of telaprevir, specifically with respect to the reported adverse effects of rash, pruritus, nausea, diarrhea, vomiting, anal or rectal discomfort (including hemorrhoids), dysgeusia, and fatigue. Furthermore, we will assess the incidence of anemia in the study population at weeks 1, 2, and 4.

SECONDARY OUTCOMES:
Election rate of study drug | One year
  During the study period, we will measure the proportion of health care workers who elect to take telaprevir for HCV post-exposure prophylaxis among the total number of HCW eligible to receive the study drug. We will also record the reasons why eligible HCW declined to participate in the study, if disclosed to the study staff.
Rate of HCV infection | One year
  Although this trial is not designed nor powered to study the efficacy of telaprevir for post-exposure prophylaxis, it will be important to measure the breakthrough rate of HCV in patients who elected treatment for 4 weeks and to calculate the rate of HCV among those who elect to not take telaprevir. The trial will be performed according to an intention-to-treat analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond T. Chung, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States